CLINICAL TRIAL: NCT01117857
Title: Duloxetine for Menopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Director of Clinical Services at the Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000956
Record Dates: First submitted 2010-05-03; First posted 2010-05-06 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Depression; Menopause; Vasomotor Symptoms
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): After a one-week placebo lead-in, all eligible subjects will receive Duloxetine 30 mg per day for one week. After one week on 30 mg, the dosage will be increased 60 mg Duloxetine per day for 7 weeks.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — One-week placebo lead-in, followed by Duloxetine 30 mg per day for one week. After one week on 30 mg, the dosage will be increased 60 mg per day for the remaining 7 weeks of the study.
  Other Names: Cymbalta

SUMMARY:
The primary objective of the study is to determine if an eight-week intervention with duloxetine significantly reduces depressive symptoms in symptomatic menopausal women. It is hypothesized that an eight-week trial with duloxetine promotes significant improvement in depression symptoms in menopausal women. The secondary aim of the study is to examine if an eight-week intervention with duloxetine significantly reduces vasomotor symptoms in symptomatic menopausal women. It is hypothesized that an eight-week trial with duloxetine promotes significant improvement in vasomotor symptoms in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women age 40 years old or older
* Menopausal symptoms of at least 3 months duration, including irregular periods and/or hot flushes
* Minimum score of 15 on the Hamilton Rating Scale for Depression (17-item),
* Patients will meet criteria for a major depressive episode, verified using the Mini International Neuropsychiatric Interview (MINI).
* Subjects will be able to be treated on an outpatient basis, and
* Subjects will be able to provide written informed consent

Exclusion Criteria:

* Subjects presently taking antidepressant medication,
* Subjects currently using hormone replacement therapy,
* Other Axis I disorders, except Generalized Anxiety Disorder or Panic Disorder, according to the Mini International Neuropsychiatric Interview (MINI)
* "uncontrolled" narrow angle glaucoma
* known hypersensitivity to duloxetine or any of the inactive ingredients
* treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or potential need to use an MAOI during the study or within 5 days of discontinuation of study drug.
* Presence of psychotic symptoms,
* History of mania or hypomania,
* HAM-D suicide item score > 3,
* End stage renal disease or severe renal impairment
* Abnormal uterine bleeding (heavy or prolonged uterine bleeding, menstrual periods occurring more frequently than every 3 weeks, bleeding after sexual intercourse, spotting between periods) that has not been evaluated by a gynecologist.
* Subjects with serious or unstable medical illness, including alcohol or substance abuse, cardiovascular, hepatic, respiratory, endocrine, neuralgic, or hematologic disease, history of seizure disorder
* Subjects taking medications that may interact with duloxetine

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Freeman MP, Hirschberg AM, Wang B, Petrillo LF, Connors S, Regan S, Joffe H, Cohen LS. Duloxetine for major depressive disorder and daytime and nighttime hot flashes associated with the menopausal transition. Maturitas. 2013 Jun;75(2):170-4. doi: 10.1016/j.maturitas.2013.03.007. Epub 2013 Apr 17. PMID 23602542
- See also: Related Info — http://www.womensmentalhealth.org/clinical-and-research-programs/registry-signup/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 29 subjects consented, 7 were found to be ineligible at the screening visit.
Period: Overall Study
Arm/Group | Duloxetine
Started | 22
Completed | 13
Not Completed | 9
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Of 29 subjects who consented, 7 were ineligible at the screening visit. Out of the 22 remaining subjects, 19 received study medication.
Arm/Group | Duloxetine
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Marital Status [Number; unit: participants]
  Married | 3
  Separated/divorced/widowed | 5
  Never married/single | 8
  Decline to answer | 3
Education [Number; unit: participants]
  Less than high school degree | 1
  High school diploma or GED | 5
  Some college | 9
  Bachelor's degree | 4
Employment Status [Number; unit: participants]
  Full- or part-time work | 4
  Homemaker | 4
  Unemployed/disabled | 7
  Student | 1
  Volunteer | 1
  Retired | 2
Menopause Status [Number; unit: participants]
  Perimenopausal | 11
  Naturally Postmenopausal | 7
  Surgically Postmenopausal | 1
Past hormone therapy use [Number; unit: participants]
  Yes | 1
  No | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Scores as Measured by the Hamilton Rating Scale for Depression
Description: The HAM-D is a 17-item well-validated and reliable measure of current depressive symptoms and their severity. Eight items are scored on a five-point scale (0-4), and nine are scored on a three-point scale (0-2) for a total score range of 0-50. A higher score indicates greater symptom severity.
Time Frame: Baseline to week 9
Population: Of the 19 participants who received study medication, 16 were considered evaluable for the purpose of analyses as they returned for at least one assessment after starting the study intervention.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 16
units on a scale | -7.5 [-11 to -4]

2. Secondary Outcome: Change in Menopause Symptoms as Measured by the Greene Climacteric Scale
Description: The Greene Climacteric Scale (GCS) is a 21-item scale used to quantify the severity of perimenopausal somatic symptoms. Each item is scored 0-3 for a total range of 0-63, with a higher score indicating greater symptom severity.
Time Frame: Baseline to week 9
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 16
units on a scale | -7.5 [-12.5 to -2.5]

3. Other Pre Specified Outcome: Change in Anxiety as Measured by the Generalized Anxiety Disorder Questionnaire (GAD-7)
Description: The GAD-7 is a valid and efficient tool for screening anxiety and assessing its severity in clinical practice and research. Subjects rate the items for severity on a 4-point scale from 0 (not at all) to 3 (nearly every day) for a total range of 0-21. A higher score indicates greater anxiety symptom burden.
Time Frame: Baseline to week 9
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 16
units on a scale | -2.5 [-7.5 to -0.5]

4. Other Pre Specified Outcome: Change in Hot Flash Interference With Daily Activities and Quality of Life as Measured by the Hot Flash Related Daily Interference Scale (HFRDIS)
Description: The HFRDIS is a 10-item self-report questionnaire in which subjects rate the degree to which hot flashes interfere with daily activities and quality-of-life during the prior week. Each item is rated on a scale from 0 (does not interfere) to 10 (completely interferes) for a total score range of 0-100 (higher score indicates greater symptom burden/interference).
Time Frame: Baseline to week 9
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 16
units on a scale | -13.5 [-44 to -7]

5. Other Pre Specified Outcome: Change in Overall Well Being Measured by the Clinical Global Impression Scale (CGI)
Description: The CGI is a scale to measure the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Severity is ranked 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. A higher score indicates greater symptom severity.
Time Frame: Baseline to week 9
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 16
units on a scale | -2 [-3 to -1]

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 9/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine (N=22)
Dry Mouth (Gastrointestinal disorders) | 5
Gastrointestinal Discomfort (Gastrointestinal disorders) | 7
Muscle tension and aches (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No